CLINICAL TRIAL: NCT07196605
Title: Efficacy and Safety of Sodium Sivelestat as an Adjunct to Mechanical Thrombectomy in Acute Large Vessel Occlusion Stroke: A Prospective Single-Arm Exploratory Study
Brief Title: Sodium Sivelestat With Mechanical Thrombectomy for Acute Stroke: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAT-TOP 2
Record Dates: First submitted 2025-09-21; First posted 2025-09-29 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke; Neutrophil Extracellular Traps Formation; Large Vessel Occlusion; Thrombectomy
Keywords: Endovascular Thrombectomy; Sodium sivelestat; Neutrophil elastase
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intravenous Sodium Sivelestat Group (Experimental): For enrolled patients, administer intravenous sodium sivelestat as soon as possible (recommended within 2 hours). The daily dosage is 4.8 mg/kg, delivered via continuous infusion with a microinfusion pump or intravenous drip, for a total duration of 5 days.
  Interventions: Drug: Sodium Sivelestat

INTERVENTIONS:
Drug: Sodium Sivelestat — For enrolled patients, administer intravenous sodium sivelestat as soon as possible (recommended within 2 hours). The daily dosage is 4.8 mg/kg, delivered via continuous infusion with a microinfusion pump or intravenous drip, for a total duration of 5 days

SUMMARY:
Stroke remains a major global health burden, with acute ischemic stroke (AIS) accounting for more than 65% of all cases. Endovascular thrombectomy (EVT) has been established as the standard treatment for large vessel occlusion (LVO) stroke; however, the phenomenon of "futile recanalization" remains common, with nearly half of patients failing to achieve favorable outcomes despite successful vessel reperfusion. Increasing evidence indicates that neutrophils and neutrophil extracellular traps (NETs) play pivotal roles in post-reperfusion inflammation, thrombosis, and microcirculatory dysfunction, contributing to thrombolysis resistance and poor prognosis. Neutrophil elastase (NE), a key component of NETs, exacerbates vascular injury and thrombus formation. Sodium sivelestat, a selective NE inhibitor, has demonstrated significant anti-inflammatory and organ-protective effects in patients with acute respiratory distress syndrome and in experimental models of cerebral ischemia. It can preserve blood-brain barrier integrity, attenuate brain edema, and improve neurological outcomes. Based on these findings, we propose a prospective, single-center, single-arm exploratory clinical trial to evaluate the efficacy and safety of sodium sivelestat as an adjunct to EVT in patients with acute LVO stroke within 24 hours of onset. The results of this study are expected to provide new clinical evidence for anti-inflammatory interventions aimed at reducing futile recanalization and improving functional outcomes in AIS.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms and signs consistent with focal ischemia in the anterior or posterior circulation;
2. Large vessel occlusion of the anterior or posterior circulation (internal carotid artery, M1/M2 segment of the middle cerebral artery, vertebral artery, or basilar artery) confirmed by CTA/MRA/DSA;
3. Undergoing mechanical thrombectomy;
4. Age ≥18 years, both male and female;
5. Pre-stroke modified Rankin Scale (mRS) score ≤1;
6. Time from symptom onset to thrombectomy ≤24 hours, including wake-up stroke or unwitnessed stroke; symptom onset is defined as the "last known well" (LKW);
7. National Institutes of Health Stroke Scale (NIHSS) score ≥6 at admission;
8. ASPECTS ≥3 for anterior circulation occlusion, or pc-ASPECTS ≥6 for posterior circulation occlusion;
9. Written informed consent provided by the patient or their legal representative.

Exclusion Criteria:

1. Simultaneous acute occlusion of both anterior and posterior circulation or bilateral hemispheric large vessel occlusions;
2. Complete clinical recovery at the end of EVT procedure;
3. Arterial dissection or intraoperative hemorrhage indicated by post-thrombectomy DSA;
4. Sedated and intubated patients without baseline NIHSS assessment;
5. Seizure at stroke onset interfering with baseline NIHSS assessment;
6. Bilateral fixed dilated pupils;
7. Severe allergy or absolute contraindication to sodium sivelestat;
8. Severe allergy or absolute contraindication to iodinated contrast agents;
9. Systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg, uncontrolled despite antihypertensive therapy;
10. Blood glucose <50 mg/dl (2.8 mmol/L) or >400 mg/dl (22.2 mmol/L);
11. Platelet count <50×10⁹/L;
12. Congenital or acquired bleeding diathesis, coagulation factor deficiency, or current use of oral anticoagulants with INR >1.7;
13. Severe renal impairment, defined as serum creatinine >3.0 mg/dl (265.2 μmol/L), GFR <30 ml/min, or requirement for hemodialysis/peritoneal dialysis;
14. Inability to complete 90-day follow-up (e.g., no fixed residence, overseas patient);
15. Suspected vasculitis or septic embolism;
16. Suspected aortic dissection;
17. Pre-existing neurological or psychiatric disorders interfering with stroke assessment;
18. Pregnancy or lactation;
19. Confirmed rheumatic/autoimmune disease with long-term use of immunosuppressants or corticosteroids;
20. Current treatment with chemotherapy or other immunomodulatory agents (e.g., recombinant human granulocyte colony-stimulating factor, Xuebijing, ulinastatin, etc.);
21. Participation in another clinical trial that may interfere with study outcomes;
22. Any other condition that investigators deem unsuitable for participation or that may pose significant risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportional distribution of modified Rankin Score | 90 days (±7 days) after randomization
  The mRS score range from 0 (no disability) to 6 (death)

SECONDARY OUTCOMES:
Rate of modified Rankin Scale (mRS) score of 0-1 | 90 days (±7 days) after randomization
  The mRS score range from 0 (no disability) to 6 (death)
Rate of mRS score of 0-2 | 90 days (±7 days) after randomization
  The mRS score range from 0 (no disability) to 6 (death)
Rate of mRS score of 0-3 | 90 days (±7 days) after randomization
  The mRS score range from 0 (no disability) to 6 (death)
Improvement of the National Institutes of Health Stroke Scale (NIHSS) score | 48 hours (±12 hours) after randomization
  The NIHSS score range from 0 (no deficit) to 42 (maximum deficit)
Rate of early neurological improvement | 48 hours (±12 hours) after randomization
  The NIHSS score decreased by ≥4 points compared with baseline
Improvement of the NIHSS score | 7 days (±1 days) after randomization or discharge
  The NIHSS score range from 0 (no deficit) to 42 (maximum deficit)
EQ-5D-5L | 90 days (±7 days) after randomization
  The EQ-5D 5-Levels (EQ-5D-5L) range from 5 (no problems) to 25 (extreme problems), which deceased patients have a utility of 0.
Barthel Index | 90 days (±7 days) after randomization
  The Barthel Index range from 0 (severe disability) to 100 (no disability)
Rate of intracranial hemorrhage (ICH) | Within 48 hours after randomization
  Any intracranial hemorrhage confirmed by imaging
Rate of symptomatic intracranial hemorrhage (sICH) | Within 48 hours after randomization
  The sICH was assessed based on the Heidelberg Bleeding Classification, defined as 1) ≥4 points total NIHSS at the time of diagnosis compared to immediately before worsening; 2) ≥2 point in one NIHSS category. The rationale for this is to capture new hemorrhages that produce new neurological symptoms, making them clearly symptomatic but not causing worsening in the original stroke territory; 3) Leading to intubation/hemicraniectomy/EVD placement or other major medical/surgical intervention; 4) Absence of alternative explanation for deterioration.
All-cause mortality | 90 days (±7 days) after randomization
  Death defined as a mRS score of 6

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University., Beijing, China

IPD SHARING:
Plan to Share IPD: No